CLINICAL TRIAL: NCT03106402
Title: Pseudophakic Cystoid Macular Lesions After Uncomplicated Standard Phacoemulsification
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Hong Kyun Kim, M.D, Professor, Kyungpook National University Hospital
Other Study IDs: KyungpookNUH
Record Dates: First submitted 2017-04-03; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Pseudophakic Cystoid Macular Lesions After Uncomplicated Standard Phacoemulsification

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated with topical NSAID: 197 eyes of - patients were treated with topical bromfenac sodium hydrate (Bronuck®, Taejoon Pharm. LTD.) 2times a day starting 1 day before surgery and continued for 2 weeks after surgery.
  Interventions: Drug: topical bromfenac sodium hydrate
- Treated without topical NSAID: 147 eyes did not receive topical NSAID after cataract surgery

INTERVENTIONS:
Drug: topical bromfenac sodium hydrate
  Groups: Treated with topical NSAID

SUMMARY:
To assess the incidence, risk factors and clinical courses of cystic macular lesions (CMLs) after uncomplicated phacoemulsification and evaluate the efficacy of topical NSAIDs on the prevention of pseudophakic cystic macular lesions

DETAILED DESCRIPTION:
344 Patients undergoing uncomplicated standard phacoemulsification at Kyungpook National University Hospital from 2013 to 2015 were reviewed. CMLs, which is any cystic fluid collections after cataract surgery, were confirmed by preoperative and postoperative optical coherence tomography(OCT) on preoperative, postoperative 1month and 3months examinations. CMLs were classified into two groups: cystic macular edema(CME) and microcystic macular edema(MME).

ELIGIBILITY:
Inclusion Criteria:

* patients who had phacoemulsification and were treated postoperatively at the Kyungpook National University Hospital, Daegu, Korea, from Oct 2013 to June 2015.

Exclusion Criteria:

* patients had complicated cataract surgery (eg, significant corneal edema, posterior capsule rupture, vitreous loss, dropped nuclear material, retained cortical material, or an IOL not placed in the capsular bag)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective chart review was of consecutive patients who had phacoemulsification and were treated postoperatively at the Kyungpook National University Hospital, Daegu, Korea, from Oct 2013 to June 2015.
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of CMLs | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hong Kyun Kim, M.D. PhD, Principal Investigator — Kyungpook National University Hospital

IPD SHARING:
Plan to Share IPD: Undecided